CLINICAL TRIAL: NCT06136975
Title: The Efficacy of Low-level Laser Therapy in Relieving Vaginal Dryness and Lower Urinary Tract Symptoms
Brief Title: Low-level Laser Therapy for Genitourinary Syndromes and Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202310054RIND
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Vaginal Atrophy; Urinary Incontinence,Stress
Keywords: Menopause; Stress urinary incontinence; Vaginal atrophy; Low-level laser therapy
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- genitourinary symptoms of menopause: Women with genitourinary symptoms of menopause (GSM). Menopause was defined as no spontaneous menstruation for at least one year. GSM defined as vulvovaginal dryness and related symptoms, such as irritation, dyspareunia, or lower urinary tract symptom (LUTS) including urinary urgency, dysuria and recurrent urinary tract infection after menopause .
  Interventions: Device: Low-level laser therapy
- stress urinary incontinence: Women with stress urinary incontinence (SUI). SUI was defined as involuntary loss of urine on effort or physical exertion including sporting activities, or on sneezing or coughing.
  Interventions: Device: Low-level laser therapy

INTERVENTIONS:
Device: Low-level laser therapy — The treatment was once a week for eight weeks. The patient was in a supine position. The gain medium of the laser was Gallium-Aluminum-Arsenide. The laser was introduced into vagina via a silicon vaginal probe inserted by a doctor for 30 minutes (wavelength 660nm, power density 18.17mW/cm2, energy density 0.018J/cm2s, total energy density 32.4J/cm2).

SUMMARY:
Genitourinary syndrome of menopause (GSM) and stress urinary incontinence (SUI) are common for women. Low-level laser therapy (LLLT) was applied for wound healing, but there was no study regarding treatment effect of GSM and SUI. This retrospective study aims to assess the efficacy of LLLT in alleviating GSM and SUI.

DETAILED DESCRIPTION:
Between September 2022 and August 2023, all women who received LLLT for GSM and SUI at the gynecologic outpatient clinic of a hospital were retrospectively reviewed. The treatment was once a week for eight weeks. Vaginal health index (VHI) and questionnaires before and after treatment for evaluation of lower urinary tract symptoms (LUTS) and quality of life are the outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* women with GSM and SUI
* Received LLLT at the gynecologic outpatient clinic

Exclusion Criteria:

* More or equal to stage 2 pelvic organ prolapse defined by pelvic organ prolapse-quantification system
* Ongoing urinary tract infection or vaginitis with the pathogen in the previous 2 weeks
* Bladder calculus
* Neurogenic bladder due to radical hysterectomy or injury of the central nervous system
* A preexisting malignant pelvic tumor.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The consecutive women who received LLLT at the gynecologic outpatient clinic were retrospectively reviewed. Menopause was defined as no spontaneous menstruation for at least one year. GSM is defined as vulvovaginal dryness and related symptoms, such as irritation, dyspareunia, or lower urinary tract symptoms (LUTS) including urinary urgency, dysuria, and recurrent urinary tract infection after menopause. SUI was defined as involuntary loss of urine on effort or physical exertion including sporting activities, or on sneezing or coughing.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Vaginal health | 8 weeks
  Vaginal health index, each of these 5 items is evaluated by means of a scale from 1 (none) to 5 (excellent) and then the average of the scores is calculated. A value of ≤15 (= cut-off) is generally considered for the diagnosis of low vaginal health.

SECONDARY OUTCOMES:
Urinary incontinence | 8 weeks
  ICIQ-SF: International Consultation on Incontinence Questionnaire - Short Form. Scoring scale: 0-21. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-chi Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Pei-chi Wu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets analyzed during the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Phillips NA, Bachmann GA. The genitourinary syndrome of menopause. Menopause. 2021 Feb 1;28(5):579-588. doi: 10.1097/GME.0000000000001728. PMID 33534428
- [Result] Gambacciani M, Palacios S. Laser therapy for the restoration of vaginal function. Maturitas. 2017 May;99:10-15. doi: 10.1016/j.maturitas.2017.01.012. Epub 2017 Feb 4. PMID 28364861
- [Result] Long CY, Wu PC, Chen HS, Lin KL, Loo Z, Liu Y, Wu CH. Changes in sexual function and vaginal topography using transperineal ultrasound after vaginal laser treatment for women with stress urinary incontinence. Sci Rep. 2022 Mar 2;12(1):3435. doi: 10.1038/s41598-022-06601-0. PMID 35236871
- [Result] Rola P, Doroszko A, Derkacz A. The Use of Low-Level Energy Laser Radiation in Basic and Clinical Research. Adv Clin Exp Med. 2014 September-October;23(5):835-842. doi: 10.17219/acem/37263. PMID 25491701
- [Result] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Result] Palacios S. Assessing symptomatic vulvar, vaginal, and lower urinary tract atrophy. Climacteric. 2019 Aug;22(4):348-351. doi: 10.1080/13697137.2019.1600499. PMID 31157569
- [Result] Huang L, Zhang SW, Wu SL, Ma L, Deng XH. The Chinese version of ICIQ: a useful tool in clinical practice and research on urinary incontinence. Neurourol Urodyn. 2008;27(6):522-4. doi: 10.1002/nau.20546. PMID 18351586